CLINICAL TRIAL: NCT03606954
Title: Evaluation of Topical Corticosteroids Potency in Combination Preparations in Healthy Volunteers
Brief Title: Potency of Topical Corticosteroids in Combination Preparations
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ben-Gurion University of the Negev (Other)
Collaborators: Soroka University Medical Center (Other)
Responsible Party: Principal Investigator, Alex Zvulunov, Head, Department of Dermatology, Ben-Gurion University of the Negev
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 0316-17-SOR
Record Dates: First submitted 2018-07-21; First posted 2018-07-31 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Skin Toxicity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: double-blind controlled comparative study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combination topical corticosteroid (Active Comparator): The combination topical corticosteroid will be applied to specific and marked sites on the forearms (on the flexor side of the forearm- 5*5 cm with a distance of 3 cm) - two sites on both forearms of every subject (4 sites in total). The nature of this application method will enable the measurement of the level of potency of each drug, in a manner that is comparative, neutralizing thus the influence of inter-subject variability.
  The drugs will be topically applied (50 microliter on each site) for 16 hours, utilizing an occlusive dressing bandage such as Tegaderm. The vasoconstriction test will be preformed both before and after drug application. The vasoconstriction in each subject will be graded on the Olsen scale
  Interventions: Combination Product: Combination topical corticosteroid
- Non-combination topical corticosteroid (Active Comparator): The non-combination topical corticosteroid will be applied to specific and marked sites on the forearms (on the flexor side of the forearm- 5*5 cm with a distance of 3 cm) - two sites on both forearms of every subject (4 sites in total). The nature of this application method will enable the measurement of the level of potency of each drug, in a manner that is comparative, neutralizing thus the influence of inter-subject variability.
  The drugs will be topically applied (50 microliter on each site) for 16 hours, utilizing an occlusive dressing bandage such as Tegaderm. The vasoconstriction test will be preformed both before and after drug application. The vasoconstriction in each subject will be graded on the Olsen scale
  Interventions: Combination Product: Combination topical corticosteroid

INTERVENTIONS:
Combination Product: Combination topical corticosteroid — Comparison of a vasoconstriction index between the 2 study arms

SUMMARY:
Several combination topical drugs are available on the market. The potency of corticosteroids depends on a particular molecular structure and the skin penetration properties. Besides molecular structure, a penetration of a corticosteroid molecule correlates with physical properties of the vehicle which depend on physical properties of the vehicle constituents.

Vasoconstriction assay is considered as the gold standard for testing potency of topical corticosteroids.

DETAILED DESCRIPTION:
Primary outcome: Change in Vasoconstriction index following application of topical corticosteroids that are incorporated with or without an antibiotic and/or antifungal drugs in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* No prior history of internal diseases that required vaccine-suppressing treatments
* Absence of an active skin disease.

Exclusion Criteria:

* Treatment with topical corticosteroids in the 4 weeks prior to the study
* Immune-suppressive treatment in the 4 weeks prior to the study
* Pregnancy or breast feeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-11 (Estimated); Primary Completion 2019-03 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Vasoconstriction Index (VI) measured by Skin Color Reflectometry | 24 hours
  VI change following application topical corticosteroids that are incorporated with an antibiotic and/or antifungal drugs.

CONTACTS AND LOCATIONS:
Overall Officials: Raed Khoury, MD, Principal Investigator — Soroka University Medical Center & Ben Gurion University

IPD SHARING:
Plan to Share IPD: Undecided